CLINICAL TRIAL: NCT01286363
Title: Preferred Chewing Side, Symmetry of Bite Force and Occlusal Contact Area of Subjects With Different Craniofacial Vertical Dimensions
Brief Title: Facial Patterns and Masticatory Symmetries
Status: Completed | Type: Observational
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Renata Cunha Matheus Rodrigues Garcia, Piracicaba Dental Schoo, State University of Campinas
Other Study IDs: monegfg11
Record Dates: First submitted 2011-01-24; First posted 2011-01-31 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Facies
Keywords: Bite force; Dental occlusion; Face; Mastication; Morphology
MeSH Terms: conditions — Facies; Bites and Stings

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Brachyfacial: Subjects with a horizontal facial growth pattern
- Mesofacial: Subjects with a balanced facial growth pattern
- Dolichofacial: Subjects with a vertical facial growth pattern

SUMMARY:
The purpose of this study is to evaluate chewing side preference, and lateral asymmetry of occlusal contact area and bite force of individuals with different craniofacial patterns

DETAILED DESCRIPTION:
Dolichofacial subjects presents poorer mechanical advantage, less efficiency in masticatory muscles during mastication and in generating bite force, smaller occlusal contact area and masticatory capacity when compared to brachyfacial individuals.

Wide, bilateral chewing cycles were related to better masticatory performance, however, unilateral chewing was reported to be very common in population, and it has been associated to lateral asymmetry on bite force and occlusal contact area.

It has been reported that dolichofacial subjects need greater muscular effort during mastication when compared to meso and brachyfacial subjects. This may cause functional overloading of weaker masticatory muscles, and may lead to functional asymmetries.

ELIGIBILITY:
Inclusion Criteria:

* Full dentition, good general and oral health

Exclusion Criteria:

* Facial deformities
* Severe malocclusion
* History of signs and symptoms of temporomandibular disorder
* History of parafunctions
* History of maxillofacial surgery or jaw injuries and orthodontic treatment concluded in the last 2 years

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Students and staff of Piracicaba Dental School, and individuals seeking for dental treatment at the same institution
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2006-09; Primary Completion 2007-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Masticatory movements during mastication | 2 hours
  A jaw tracking device was positioned on subjects face, who were asked to chew an artificial material in their habitual way. Tracings of jaw lateral movements during mastication were analyzed to classify in which side each chewing stroke was taken. If 80 percent or more chewing cycles were classified as left or right, the subjects were considered as unilateral chewer.

SECONDARY OUTCOMES:
Bite force and occlusal contact area | 2 hours
  A strain gauge was positioned on subject's first molar region unilaterally to measure the symmetry of bite force. The individual was asked to bite as hard as possible. The procedure was repeated to the other side, and the bite symmetry of sides was analyzed.
  To evaluate symmetry of occlusal contact area, a registration of posterior teeth was performed with the subjects in maximal intercuspal position. The registration was digitalized, discolored, color inverted and adjusted for size to evaluate thickness of registration material using a software.

CONTACTS AND LOCATIONS:
Overall Officials: Simone G Farias Gomes, PhD, Principal Investigator — Universidade Federal de Pernambuco; William Custodio, MS, Study Chair — Piracicaba Denal School, State University of Campinas; Fernanda Faot, PhD, Study Chair — Federal University of Pelotas; Altair A Del Bel Cury, PhD, Study Director — Piracicaba Dental School, State University of Campinas; Renata CM Rodrigues Garcia, PhD, Study Director — Piracicaba Dental School, State University of Campinas
Locations (1):
- Piracicaba Dental School, Piracicaba, São Paulo, Brazil

REFERENCES:
- [Background] Gomes SG, Custodio W, Faot F, Del Bel Cury AA, Garcia RC. Masticatory features, EMG activity and muscle effort of subjects with different facial patterns. J Oral Rehabil. 2010 Nov;37(11):813-9. doi: 10.1111/j.1365-2842.2010.02075.x. Epub 2010 Aug 19. PMID 20726943
- [Background] Martinez-Gomis J, Lujan-Climent M, Palau S, Bizar J, Salsench J, Peraire M. Relationship between chewing side preference and handedness and lateral asymmetry of peripheral factors. Arch Oral Biol. 2009 Feb;54(2):101-7. doi: 10.1016/j.archoralbio.2008.09.006. Epub 2008 Oct 22. PMID 18947820
- [Background] Garcia-Morales P, Buschang PH, Throckmorton GS, English JD. Maximum bite force, muscle efficiency and mechanical advantage in children with vertical growth patterns. Eur J Orthod. 2003 Jun;25(3):265-72. doi: 10.1093/ejo/25.3.265. PMID 12831216
- [Background] Sonnesen L, Bakke M, Solow B. Temporomandibular disorders in relation to craniofacial dimensions, head posture and bite force in children selected for orthodontic treatment. Eur J Orthod. 2001 Apr;23(2):179-92. doi: 10.1093/ejo/23.2.179. PMID 11398555
- [Derived] Gomes SG, Custodio W, Faot F, Cury AA, Garcia RC. Chewing side, bite force symmetry, and occlusal contact area of subjects with different facial vertical patterns. Braz Oral Res. 2011 Sep-Oct;25(5):446-52. doi: 10.1590/s1806-83242011005000014. PMID 22031059